CLINICAL TRIAL: NCT05541211
Title: Comparing the Effects of Coeliac Plexus Neurolysis Versus Splanchnic Nerve Neurolysis for Non-pancreatic Upper Intra-abdominal Cancer Pain: a Prospective Randomized Study
Brief Title: Coeliac Plexus Neurolysis Versus Splanchnic Nerve Neurolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Honorary Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW22-536
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: The randomization sequence will be generated by Microsoft Excel software. Blocked randomization will be done with an allocation ratio of 1:1. This will be prepared by a statistician unaware of the nature of the clinical study. The sequence will be concealed in opaque envelopes and opened by an investigator just before the procedure. The patients and independent investigators collecting outcome data will be blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients and independent investigators collecting outcome data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coeliac plexus neurolysis (CPN) (Active Comparator): Coeliac plexus neurolysis (CPN) will be performed bilaterally. Neurolytic solution will be injected around the coeliac plexus (a network of nerves located in the abdomen).
  Interventions: Other: Coeliac plexus neurolysis
- Splanchnic nerve neurolysis (SNN) (Experimental): Splanchnic nerve neurolysis (SNN) will be performed bilaterally. Neurolytic solution will be injected around the splanchnic nerves (a nerve located at thoracic trunk).
  Interventions: Other: Splanchnic nerve neurolysis

INTERVENTIONS:
Other: Coeliac plexus neurolysis — Coeliac plexus neurolysis (CPN) will be performed bilaterally. Neurolytic solution will be injected around the coeliac plexus (a network of nerves located in the abdomen).
  Arms: Coeliac plexus neurolysis (CPN)
Other: Splanchnic nerve neurolysis — Splanchnic nerve neurolysis (SNN) will be performed bilaterally. Neurolytic solution will be injected around the splanchnic nerves (a nerve located at thoracic trunk).
  Arms: Splanchnic nerve neurolysis (SNN)

SUMMARY:
Pain is prevalent among patients with gastrointestinal cancers. Standard procedures such as coeliac plexus neurolysis (CPN) is effective in reducing pain, opioid requirement and related side effects for pancreatic cancer cases. Meanwhile, splanchnic nerve neurolysis (SNN) as an alternative to CPN is more effective for cancer pain relief.

Although previous studies investigating the role of CPN/SNN mainly focus on pancreatic cancer cases, their efficacy on non-pancreatic abdominal cancer pain may not be accurately determined.

DETAILED DESCRIPTION:
Pain is prevalent among patients with gastrointestinal cancers. There is abundant evidence that coeliac plexus neurolysis (CPN) is effective in reducing pain, opioid requirement and related side effects for pancreatic cancer cases while the evidence for other upper abdominal cancer pain is less robust but emerging. Meanwhile, there is an increasing interest in utilising splanchnic nerve neurolysis (SNN) as an alternative to CPN for cancer pain relief.

Although previous studies investigating the role of CPN/SNN involved heterogenous types of intra-abdominal malignancies, majority of cases were pancreatic cancer. Therefore, their efficacy on non-pancreatic abdominal cancer pain may not be accurately determined.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Diagnosis of unresectable intra-abdominal cancer
* Visceral pain attributable to the cancer with NRS >= 4
* Able to understand instructions, give consent, complete questionnaires

Exclusion Criteria:

* Primary pancreatic cancer or metastatic disease involving pancreas
* Gross celiac axis distortion identified on imaging
* Acute abdomen condition eg. Intraabdominal sepsis, tumor rupture
* Other non-cancer causes attributable to the pain
* Gross ascites
* Previous coeliac plexus or splanchnic nerve neurolysis
* Contraindications to neurolytic procedures eg. Bleeding tendency; local or systemic infections; allergic to local anesthetics, contrast or alcohol; intestinal obstruction; anatomical distortion along needle trajectory
* Patients believed to be inappropriate for study by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
pain score | at one week after procedure
  Pain intensity using numerical rating scale from 0 to 10 where 0 is no pain and 10 is the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No